CLINICAL TRIAL: NCT03744520
Title: Assessment of Dermatomal Sensorial Block of Erector Spinae Plane Block: Randomized, Prospective, Study
Brief Title: Sensorial Block Assessment of Erector Spinae Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Onur Selvi (Other)
Responsible Party: Sponsor-Investigator, Onur Selvi, MD, Maltepe University
Organization: Maltepe University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Sensorial Block assessment
Record Dates: First submitted 2018-10-25; First posted 2018-11-16 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Regional Anesthesia Morbidity
Keywords: regional anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ESP block group (Experimental): The patients who had paravertebral interfacial plane block for postoperative analgesia
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — Local anesthetic infiltration is applied between the erector spinae muscle fascia and transverse process.

SUMMARY:
Ultrasound-guided erector spinae plane blocks are used as postoperative analgesia method for abdominal, chest and hip surgeries. Regional techniques are well-described methods for postoperative analgesia. However, the sensorial dermatomal spread of regional block varies depending on the multiple variables as the level of the block, local analgesic concentration etc. The aim of this study is to observe dermatomal evaluation of sensorial block.

ELIGIBILITY:
Inclusion Criteria:

* The patients who received successful erector spinae plane block for postoperative analgesia

Exclusion Criteria:

* Patients under 18 years old
* Patients who are not able to communicate with
* Patients who are on medication which may change the perception of pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

PRIMARY OUTCOMES:
Spread of sensorial block | in postoperative sixth hours
  The sensorial block will be evaluated with dermatomal examination

CONTACTS AND LOCATIONS:
Locations (1):
- Maltepe University Medical Faculty, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No